CLINICAL TRIAL: NCT06947980
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Phase 2 Study to Evaluate the Efficacy and Safety of CM512 in Patients With Moderate-to-Severe Atopic Dermatitis
Brief Title: Study of CM512 in Patients With Moderate-to-Severe Atopic Dermatitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CM512-101102
Record Dates: First submitted 2025-04-25; First posted 2025-04-27 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (Placebo Comparator)
  Interventions: Drug: Placebo Comparator
- Group 2 (Experimental)
  Interventions: Biological: CM512
- Group 3 (Experimental)
  Interventions: Biological: CM512
- Group 4 (Experimental)
  Interventions: Biological: CM512
- Group 5 (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Placebo Comparator — Placebo subcutaneous injection
  Arms: Group 1; Group 5
Biological: CM512 — CM512 subcutaneous injection
  Arms: Group 2; Group 3; Group 4

SUMMARY:
A Phase 2 study designed to evaluate the efficacy and safety of CM512 in adult patients with moderate-to-severe Atopic Dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of AD for at least 1 year according to the American Academy of Dermatology's consensus criteria prior to the screening visit meeting all of the following criteria:
* EASI≥16 at Screening and Baseline visits;
* Investigator's Global Assessment (IGA) score of≥3 at Screening and Baseline visits;

  * 10% Body Surface Area (BSA) of AD involvement at Screening and Baseline visits;
* Mean of weekly Pruritus Numeric Rating Scale (NRS) severity score≥4 at Baseline;

Exclusion Criteria:

* Not enough washing-out period for previous therapy.
* Concurrent disease/status which may potentially affect the efficacy/safety judgement.
* Organ dysfunction.
* Pregnancy.
* Other.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-19 (Actual); Primary Completion 2026-07-18 (Estimated); Study Completion 2026-11-07 (Estimated)

PRIMARY OUTCOMES:
Percent change from Baseline in Eczema Area and Severity Index (EASI) at Week 24 | Baseline, Week 24
  The EASI score is used to measure the severity and extent of AD and measured erythema, edema/papulation, excoriation and lichenification on 4 anatomic regions of the body: head and neck, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Zhang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No